CLINICAL TRIAL: NCT03844607
Title: Combined tDCS and Cognitive Training to Reduce Impulsivity in Patients With Traumatic Brain Injury
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Minneapolis Veterans Affairs Medical Center (U.S. Federal Agency)
Collaborators: Minnesota Office of Higher Education (Other Government); Center for Veterans Research and Education (Other); The Defense and Veterans Brain Injury Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Casey Gilmore, PhD, Research Scientist, Minneapolis Veterans Affairs Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: VAM-18-00308
Record Dates: First submitted 2019-02-13; First posted 2019-02-18 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Traumatic Brain Injury; Impulsivity
MeSH Terms: conditions — Brain Injuries, Traumatic; Impulsive Behavior

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Active tDCS (Experimental): Participants will receive 5 sessions of cognitive training concurrent with transcranial direct current stimulation (anode over left frontal cortex, cathode over right frontal cortex; 2 mAmps for 20 minutes).
  Interventions: Device: Active Transcranial Direct Current Stimulation (tDCS)
- Sham tDCS (Sham Comparator): Participants will receive 5 sessions of cognitive training concurrent with sham tDCS. For sham tDCS, electrodes are placed at the same locations as for active tDCS, but current is ramped up for the initial 30 secs, then immediately ramped back down. This method mimics the initial physical sensation of stimulation, but there is no active current for the remainder of the session.
  Interventions: Device: Sham Transcranial Direct Current Stimulation (tDCS)

INTERVENTIONS:
Device: Active Transcranial Direct Current Stimulation (tDCS) — Cognitive training concurrent with 2 mAmps of anodal stimulation applied to the left frontal cortex for 20 minutes.
  Arms: Active tDCS
Device: Sham Transcranial Direct Current Stimulation (tDCS) — Cognitive training concurrent with sham tDCS (30 secs ramp up/ramp down of current at beginning of session).
  Arms: Sham tDCS

SUMMARY:
Behavioral changes following a traumatic brain injury (TBI) are one of the biggest challenges for patients, as well as their family members and others involved in their recovery. One of the most common behavioral changes following TBI is the emergence of impulsive behavior, which has been associated with destructive, suicidal, and aggressive behavior, and is related to poor rehabilitation program adherence. The primary objective of this study is to investigate the effect of a novel neuroplasticity based intervention that combines cognitive training and transcranial direct current stimulation (tDCS) to reduce impulsivity and to improve outcomes and quality of life for those who have suffered a TBI.

DETAILED DESCRIPTION:
Behavioral changes following a traumatic brain injury (TBI) are one of the biggest challenges for patients, as well as their family members and others involved in their recovery. One of the most common behavioral changes following TBI is the emergence of impulsive behavior, which has been associated with destructive, suicidal, and aggressive behavior, and is related to poor rehabilitation program adherence. The primary objective of this study is to investigate the effect of a novel neuroplasticity based intervention approach utilizing transcranial direct current stimulation (tDCS) to alter brain neuroplasticity combined with cognitive training tasks selected to functionally target cognition and brain circuits that are impaired in those TBI patients with impulsive behavior.

This double-blind, randomized, placebo (sham) controlled study will recruit 30 Veterans with a history of mild, moderate or severe TBI, who exhibit a variety of impulsive behaviors. Participants will be randomly assigned to receive either active or sham tDCS, both paired with cognitive training tasks, once a day for five days. Additionally, participants will attend three follow up visits at 1, 2, and 3 months after the course of intervention visits is completed. Functional magnetic resonance imaging (fMRI) will be collected before and after intervention, to measure brain activity changes across time depending on intervention type.

ELIGIBILITY:
Inclusion Criteria:

Participants will be included in the study if they:

* have a clinical history of impulsive behavior, including substance abuse, gambling problems, legal issues such as DUI, violent acts, aggression, history of suicidality, or ADHD as assessed by the patient's clinical provider and/or screen of medical records
* are age 18 or older
* are receiving services from the Minneapolis VA Health Care System
* are stable on any medications for at least 1 week at the baseline visit
* have a diagnosis of mild, moderate, or severe TBI (as defined by VA/DoD Clinical Practice Guidelines criteria)

Exclusion Criteria:

Persons will be excluded from this study if they:

* have a significant neurological disorder based on the Principal Investigators judgment that would impact risk
* diagnosed with current active psychosis or mania
* have metallic cranial plates/screws or implanted devices
* have eczema on scalp or other scalp lesions or skin disorders that may become irritated by stimulation
* are pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2019-01-08 (Actual); Primary Completion 2023-03-16 (Actual); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
Change in Barratt Impulsiveness Scale (BIS) | Change between baseline and 1 week follow-up; 1, 2, and 3 months following intervention
  Differences in magnitude of change in BIS scores between active tDCS and sham groups from baseline to follow-up sessions. Higher total score on the BIS indicates higher levels of impulsivity.

SECONDARY OUTCOMES:
Change in choice of higher risk option in the Risk Task | Change between baseline and 1 week follow-up; 1, 2, and 3 months following intervention
  Differences in magnitude of change in choice of higher risk option during the Risk Task between active tDCS and sham groups from baseline to follow-up sessions. Greater choice of higher risk options in the Risk Task indicates higher levels of risk-taking and impulsivity.
Change in Brain Functional Connectivity as measured by functional magnetic resonance imaging (fMRI) | Change between baseline and 1 week follow-up
  Compare magnitude of change in frontal-striatal functional connectivity between active tDCS and sham groups from baseline to following the 5 sessions of intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- Minneapolis VA Medical Center, Minneapolis, Minnesota, United States